CLINICAL TRIAL: NCT02176941
Title: Short Telomere in Patients at High Cardiovascular Risk: a Simple Marker or a Major Determinant of Accelerated Arterial Aging
Brief Title: Telomeres and Arterial Aging
Acronym: TELARTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: National Research Agency, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Assistance Publique Hopitaux De Marseille (Other); University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A00298-39
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Atherosclerotic Disease
Keywords: Telomere Length; Arterial Aging; Endothelial Progenitor Cells; Inflammation; Atherosclerosis
MeSH Terms: conditions — Inflammation; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skeletal Muscle, skin, fat (as surgical waste) and Blood sampling DNA extractions and telomere length measurements (Southern) in muscular cells, white blood cells and endothelial progenitor cells.
  Determination, isolation and characterization of endothelial progenitor cells Microparticle (MP) von Willebrand Factor : vWF, CD146, CD31 Tissue plasminogen activator/plasminogen activator inhibitor-1 complexes thrombomodulin, endothelial protein C receptor, free tissue factor pathway inhibitor sirtuin proteins Biological phenotyping of inflammatory factors in plasma : IL2, IL4, IL6, IL8, IL10, VEGF, IFNG, TNFA, IL1A, IL1B, MCP1, EGF, CRP, Haptoglobine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ATHEROMA group: "ATHEROMA" group will include patients undergoing cardiovascular surgery or have pacemaker/defibrillator implantation and have a clinically significant atherosclerotic disease
- Control Surgery group: "Control Surgery" group will include patients undergoing other surgery or pacemaker/defibrillator implantation without evidence of clinical CV disease or history of previous CV disease.

SUMMARY:
The prevailing view in telomere epidemiology is that leukocyte telomere length (LTL) is associated with atherosclerosis and accelerated aging since it serves as a biomarker of the cumulative burden of inflammation and oxidative stress during adult life. Our recent results however, indicate that telomere length (TL) is mainly determined at birth and childhood. Since short telomeres ante cede atherosclerosis, the investigators hypothesize that TL is not just a simple marker, but a real determinant of arterial aging. That is because TL reflects cellular repair capacity and a short LTL denotes diminished repair reserves. This hypothesis cannot be tested by measurements of LTL alone, since this parameter reflects TL at birth and its age-dependent attrition thereafter. The investigators propose, therefore, a model that makes it possible to examine different elements of TL dynamics in different tissues: leukocytes, skeletal muscle, endothelial progenitor cells (EPCs), skin or subcutaneous fat in patients with or without atherosclerosis.

Our model is based on the following premises, which are derived from observations that TL is synchronized (equivalent) across somatic tissues/cells of the newborn:

* TL in skeletal muscle mainly reflects TL at birth
* The difference in TL between muscle and leukocytes in adults (approximately 1.5 Kbp) mainly reflects LTL attrition during the growth period, i.e., childhood/adolescence
* TL in EPCs determines the cell proliferative ability and therefore capacity for vessels repair during aging.

The general aim of the present project is to examine the links of arterial aging with TL, as expressed in different tissues, and LTL dynamics, as expressed in the difference between TLs of muscle and leukocytes.

DETAILED DESCRIPTION:
Specific objectives:

1. To determine whether TL during early development, which is primarily reflected in muscle TL, and LTL attrition during development, which is primarily expressed in the difference between muscle TL and LTL, are associated with indices of arterial aging.
2. To examine the relation between EPC-TL to endothelial regenerative capacity and endothelial function. In order to attain this objective the investigators will perform two types of experiments:

   * Measure TL in progenitor cells and relate it to clinical phenotypes of arterial aging and atherosclerosis, as well as markers of endothelial dysfunction
   * Generate in vitro progenitor cells with different TL induced by the environmental factors (oxidative stress) and assess their phenotypes concerning inflammation and microvesiculation, in order to show a possible mechanistic relationship between TL in PC and the atherogenic and the regenerative capacities of these cells.

The project is composed of 6 tasks:

T1: Recruitment and sample collection (skeletal muscle, total blood) of 170 patients with atherosclerosis and 170 controls. Performed by surgeons and cardiologists of Marseille and Nancy University hospitals T2: Characterization of arterial aging in all patients (Geriatric Dpt, Univ. hospital Nancy, Pr Benetos and AP-HM, Internal Medicine, Marseille, Dr Rossi) T3: Characterization of early and late endothelial progenitor cells (EPC): laboratory of hematology and vascular biology and in UMR_S1076 in Marseille (Prs Dignat-George and Sabatier) T4: Measurements of TL in all samples (skeletal muscle, leukocytes and EPC): UMR_S1116 Nancy (Dr Lacolley) in collaboration with Pr Aviv (University of Medicine of New Jersey) T5: Characterization of inflammation markers in blood samples: UMR_S1116 and the UMR_S1122 (Dr Siest-Visvikis, Nancy) T6: Database construction and statistical analyses (UMR_S1116)

The results of this program could completely modify the present concept on the association between TL and cardiovascular risk: Actually, if our concept of early determination of TL is valid, therefore TL could be a true determinant of the arterial aging pace, through limitation of repair capacity of cells.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged ≥ 20 years who are admitted for different types of surgery or for pacemaker/ defibrillator implantation and provide informed consent for participating in this study.

Exclusion Criteria:

Conditions which may impact telomere length:

* Patients undergoing surgery for cancer
* Patients who had had radiotherapy or chemotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited among patients admitted to the hospital either for surgery or for installing pacemakers/ defibrillators. Informed consent will be signed at the beginning of the hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Telomere Length (LT) dynamics | up to 3 years
  TL dynamics: as expressed in the difference between TLs of muscle and leukocytes.

SECONDARY OUTCOMES:
Skin telomere length | up to 3 years
Subcutaneous fat telomere length | up to 3 years

OTHER OUTCOMES:
Measure TL in progenitor cells | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Athanase BENETOS, MD, PhD, Principal Investigator — Service de Gériatrie et INSERM U1116; Université de Lorraine et CHU de Nancy; France
Locations (2):
- France (2):
  - AP Hôpitaux de Marseille, Marseille
  - Chu Nancy, Nancy

REFERENCES:
- [Derived] Lai TP, Verhulst S, Savage SA, Gadalla SM, Benetos A, Toupance S, Factor-Litvak P, Susser E, Aviv A. Buildup from birth onward of short telomeres in human hematopoietic cells. Aging Cell. 2023 Jun;22(6):e13844. doi: 10.1111/acel.13844. Epub 2023 Apr 28. PMID 37118904
- [Derived] Toupance S, Simonici S, Labat C, Dumoulin C, Lai TP, Lakomy C, Regnault V, Lacolley P, Dignat George F, Sabatier F, Aviv A, Benetos A; TELARTA consortium dagger. Number and Replating Capacity of Endothelial Colony-Forming Cells are Telomere Length Dependent: Implication for Human Atherogenesis. J Am Heart Assoc. 2021 May 18;10(10):e020606. doi: 10.1161/JAHA.120.020606. Epub 2021 May 6. PMID 33955230
- [Derived] Benetos A, Toupance S, Gautier S, Labat C, Kimura M, Rossi PM, Settembre N, Hubert J, Frimat L, Bertrand B, Boufi M, Flecher X, Sadoul N, Eschwege P, Kessler M, Tzanetakou IP, Doulamis IP, Konstantopoulos P, Tzani A, Korou M, Gkogkos A, Perreas K, Menenakos E, Samanidis G, Vasiloglou-Gkanis M, Kark JD, Malikov S, Verhulst S, Aviv A. Short Leukocyte Telomere Length Precedes Clinical Expression of Atherosclerosis: The Blood-and-Muscle Model. Circ Res. 2018 Feb 16;122(4):616-623. doi: 10.1161/CIRCRESAHA.117.311751. Epub 2017 Dec 14. PMID 29242238